CLINICAL TRIAL: NCT07236749
Title: Effect of Postoperative Oral Rinsing on Thirst-Related Discomfort, Comfort Level, and Bowel Movement in Individuals Undergoing Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Effect of Postoperative Oral Rinsing on Dehydration-Related Discomfort, Comfort, and Bowel Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Pınar YILMAZ EKER, Asst. Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-01/33
Record Dates: First submitted 2025-07-22; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Thirst; Comfort; Bowel Movements; Abdominal Surgeries
Keywords: Postoperative Thirst; Comfort; Bowel Movements; Abdominal surgeries; Nursing care; perioperative care

STUDY DESIGN:
Intervention Model Description: Randomised conrtolled trial
Who Masked: Participant
Masking Description: This study used a stratified random sampling method. Patients were stratified by clinical diagnosis and gender and randomized into blocks. Using a random number table, the first patient to arrive was assigned to the experimental group, and subsequent patients were sampled using a 1:1 allocation method until strata and blocks were equal in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal surgery patients receiving oral rinsing (Experimental): Abdominal surgery patients
  Interventions: Other: oral rinsing
- rutine service operation (Other): Abdominal surgery patients
  Interventions: Other: rutine service operation

INTERVENTIONS:
Other: oral rinsing — The experimental group received a postoperative mouth rinse with pure water.
  Arms: Abdominal surgery patients receiving oral rinsing
Other: rutine service operation — No additional intervention will be made to the control group; only data collection forms will be applied.
  Arms: rutine service operation

SUMMARY:
The aim of this study is to evaluate the effects of oral rinsing with water in the postoperative period on thirst, comfort level, and bowel motility in patients undergoing abdominal surgery under general anesthesia.

This study was conducted as a randomized controlled trial with pretest-posttest design, including intervention and control groups. It was carried out between June 2024 and December 2024 with patients undergoing elective abdominal surgery. Sample size was calculated using G*Power 3.1.9.7 software, with an effect size of 0.50, α=0.05, and power=0.85. A total of 82 participants (41 per group) were initially planned, and considering a 10% data loss, the study was completed with 98 participants (49 in each group). Patients were stratified according to their diagnoses and randomized in a 1:1 ratio using block randomization with a random number table.

Three data collection forms were used. SPSS 22.00 package program was used to analyze the data. Skewnes-Kurtosis analyses were performed to determine the conformity of the data to a normal distribution. Frequency (n) and percentage (%) distributions were calculated to determine the sociodemographic and clinical characteristics of the participants. A t-test for independent samples was used to determine the mean differences between two independent groups, a t-test for dependent samples was used to compare pre- and post-intervention measurements, and a single-factor analysis of variance (ANOVA) was used for repeated measures. Cohen's d effect size was calculated to assess the significance of the difference between the groups in terms of the intervention. Statistical significance was accepted as p<0.05.

ELIGIBILITY:
Included Criteria

* To communicate,
* Aged 18 or older,
* Agreed to participate
* Scheduled for elective surgery.

Exclusion Criteria

* Over 80 years old,
* Had a mental disorder that prevented them from rinsing their mouth,
* Unconscious after surgery, were at
* Risk of swallowing water during rinsing,
* Underwent emergency surgery.

Refusion Criteria

* Refused to complete the post-test
* Intensive care after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Scores of Mental State Assessment pre-test post-test on experimental group | 1 day
  Mini Mental State Assessment (MMSA): A cognitive screening tool with 11 items in five domains (orientation, registration, attention/calculation, recall, language). Scores range 0-30; ≤23 indicates impairment. Administration takes 5-10 minutes. Turkish validity and reliability are established.
Personal Information experimental group | 1 day
  Personal Information Form: Developed by researchers based on literature and clinical observation. The first section includes demographic and clinical data (age, gender, education, diagnosis, preoperative fasting time, postoperative oral intake time). The second section records bowel sounds.
Scores of Surgical Period Thirst Discomfort pre-test post-test on experimental group | 1 day
  Surgical Period Thirst Discomfort Scale (SPTDS): Adapted to 6 items with a 3-point Likert scale (0-2). Total score is 0-12; higher scores indicate greater thirst-related discomfort.Surgical Period Thirst Discomfort Scale (SPTDS)
Comfort levels pre-test post-test on experimental group | 1 day
  VAS-10: A 10-cm line used to evaluate comfort; 0 = lowest, 10 = highest comfort. Higher scores reflect greater comfort.
Scores of Mental State Assessment pre-test post-test on control group | 1 day
  Mini Mental State Assessment (MMSA): A cognitive screening tool with 11 items in five domains (orientation, registration, attention/calculation, recall, language). Scores range 0-30; ≤23 indicates impairment. Administration takes 5-10 minutes. Turkish validity and reliability are established.
Personal Information control group | 1 day
  Personal Information Form: Developed by researchers based on literature and clinical observation. The first section includes demographic and clinical data (age, gender, education, diagnosis, preoperative fasting time, postoperative oral intake time). The second section records bowel sounds.
Scores of Surgical Period Thirst Discomfort pre-test post-test on control group | 1 day
  Surgical Period Thirst Discomfort Scale (SPTDS): Adapted to 6 items with a 3-point Likert scale (0-2). Total score is 0-12; higher scores indicate greater thirst-related discomfort.Surgical Period Thirst Discomfort Scale (SPTDS)
Comfort levels pre-test post-test on control group | 1 day
  VAS-10: A 10-cm line used to evaluate comfort; 0 = lowest, 10 = highest comfort. Higher scores reflect greater comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar YILMAZ EKER, Asst. Prof. Dr., Principal Investigator — Cumhuriyet University; Ayşegül KAYA İMREK, Res. Asst., Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish the study in an international journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data were collected for 6 months

REFERENCES:
- [Result] Babacan-Yildiz G, Ur-Ozcelik E, Kolukisa M, Isik AT, Gursoy E, Kocaman G, Celebi A. [Validity and Reliability Studies of Modified Mini Mental State Examination (MMSE-E) For Turkish Illiterate Patients With Diagnosis of Alzheimer Disease]. Turk Psikiyatri Derg. 2016 Spring;27(1):41-6. Turkish. PMID 27369684
- [Result] Yaray O, Akesen B, Ocaklioglu G, Aydinli U. Validation of the Turkish version of the visual analog scale spine score in patients with spinal fractures. Acta Orthop Traumatol Turc. 2011;45(5):353-8. doi: 10.3944/AOTT.2011.2528. PMID 22033000
- [Result] Özsoy, H. , Güreş, Z., Dolgun, E. & Yavuz van Giersbergen, M. (2023). Cerrahi Dönem Susuzluğa Bağlı Rahatsızlık Ölçeği (CDSBRÖ) Türkçe Geçerlik ve Güvenirliği. Fırat Üniversitesi Sağlık Bilimleri Dergisi, 37 (3), 237- 242.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT07236749/Prot_SAP_ICF_000.pdf